CLINICAL TRIAL: NCT07064174
Title: Sickle Cell Kidney (SCeK) Biorepository
Brief Title: Sickle Cell Kidney Biorepository
Acronym: SCeK
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kabir Olaniran, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2022-1024
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Sickle Cell Trait; Sickle Cell Disease (SCD); Chronic Kidney Disease
MeSH Terms: conditions — Sickle Cell Trait; Anemia, Sickle Cell; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Serum, Plasma (lithium heparin and K2 EDTA), Citrate whole blood, K2EDTA Buffy coat, Urine supernatant, Urine sediment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Kidney disease is a major cause of illness and death in people with sickle cell disease and sickle cell trait. Despite these concerning facts, we do not (1) have an in-depth understanding of how kidney disease starts in sickle cell disease and sickle cell trait, (2) have detailed insights into why kidney disease is worse in people with sickle cell disease and sickle cell trait, (3) have management options that are tailored to treating or preventing kidney disease in people with sickle cell disease or sickle cell trait.

The SCeK Biorepository is a specialized, secure repository designed for the collection of blood and urine samples from people with sickle cell disease and sickle cell trait. These samples are connected to detailed medical records, with the sole purpose of allowing researchers to better understand how kidney disease starts and progresses in people with the sickle cell gene. By studying these stored samples (using new tests) together with health information, researchers can find better early warning signs of kidney injury and develop better ways to protect kidney health in people with sickle cell disease and sickle cell trait.

DETAILED DESCRIPTION:
Chronic kidney disease is one of the most common causes of morbidity and mortality in sickle cell disease, occurring at a much earlier age and with a far higher frequency as compared to the general population. Furthermore, sickle cell trait has emerged as an under-recognized major risk factor for chronic kidney disease.

Despite the seriousness of these findings, there are significant gaps in our understanding of the pathophysiology of and risk factors for incident chronic kidney disease and chronic kidney disease progression in both sickle cell disease and sickle cell trait.

The UT Southwestern and Parkland Health Sickle Cell Kidney (SCeK) Biorepository aims to address these knowledge gaps by collecting well annotated, high quality dedicated bio-samples integrated with routine clinical data to facilitate improved prognostication, provide mechanistic insights, and form the basis for the investigation of novel therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years,
2. Estimated glomerular filtration rate greater than or equal to 15 mL/min,
3. Presence of any hemoglobinopathy (will need to be confirmed by hemoglobin electrophoresis or genetic testing),
4. Controls (absence of hemoglobinopathy) will be subject to review and only selected if demographics are identical to a currently enrolled participant with a hemoglobinopathy.

Exclusion Criteria:

1. Age 66 years or older,
2. Estimated glomerular filtration rate less than 15 mL/min or on dialysis,
3. Active pregnancy (may be enrolled 4 weeks or more after delivery),
4. Active sickle cell pain episode requiring hospitalization or emergency room visit or pain infusion clinic visit (may be enrolled 2 weeks or more after resolution of severe pain),
5. Active malignancy on induction or consolidation treatment. Maintenance chemotherapy in remission will be considered,
6. Prisoners.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants include all eligible adults who are able to provide samples at the primary study site(s). Health data and surveys can be completed electronically.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2049-12 (Estimated); Study Completion 2049-12 (Estimated)

PRIMARY OUTCOMES:
Kidney function decline | 10 years
  Mean change in the estimated glomerular filtration rate per year
Albuminuria | 10 years
  Mean change in the urine albumin-to-creatinine ratio per year

SECONDARY OUTCOMES:
Mortality | 10 years
  Time to death over follow up period
Hospitalization rates | 10 years
  Frequency of hospitalizations and emergency room visits over follow up
Cardiovascular outcomes | 10 years
  Incident left ventricular hypertrophy, diastolic dysfunction, heart failure, pulmonary hypertension, or stroke.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Parkland Memorial Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be available beginning 6 months after publication of the primary results and will remain available for up to 10 years.
Access Criteria: Data will be shared with qualified researchers who provide a methodologically sound research proposal. Requests can be submitted to the study principal investigator by email. A data request portal will be added to the website in due course (www.utsouthwestern.edu/scek-study). Only researchers affiliated with academic, non-profit, or governmental institutions, pending data use agreement and ethical approval from their institutional review boards will be provided with data.